CLINICAL TRIAL: NCT04540848
Title: Post Operative Pain Control for Distal Radius Surgery: Does Exparel Injected at the Surgery Site Improve Postoperative Pain Scores at 24 and 48 Hours ?
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of ability to communicate with the study population
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Erikka L Washington, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSC-MS-20-0430
Record Dates: First submitted 2020-08-31; First posted 2020-09-07 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Post Operative Pain
Keywords: Brachial plexus block; Multimodal pain control for Distal Radius surgery; Exparel; Bupivacaine; Distal Radius Pain Control; Post operative pain Control; Supraclavicular nerve block
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Exparel plus supraclavicular block (Experimental)
  Interventions: Drug: Group A (Exparel plus supraclavicular block)
- Bupivacaine HCL plus supraclavicular block (Active Comparator)
  Interventions: Drug: Group B (Bupivacaine HCL plus supraclavicular block)
- supraclavicular block only (Active Comparator)
  Interventions: Drug: Group C(supraclavicular block only)

INTERVENTIONS:
Drug: Group A (Exparel plus supraclavicular block) — Patients will receive 20 cc (266 mg) of Exparel injected in the distal radius area and a supraclavicular block in the recovery room.The supraclavicular blocks will be ultrasound guided and consist of 20 cc of Bupivacaine HCl 0.25% .Anesthesiologist performing the block will be instructed to surround the brachial plexus with the local anesthetic, taking special care to inject in the "corner pocket".
  Arms: Exparel plus supraclavicular block
Drug: Group B (Bupivacaine HCL plus supraclavicular block) — Patients will receive 20 cc of Bupivacaine 0.25% (50mg) in the distal radius area.In the recovery room the patient will be given the supraclavicular block which will be ultrasound guided and consisting of 20 cc of Bupivacaine HCl 0.25% .Anesthesiologist performing the block will be instructed to surround the brachial plexus with the local anesthetic, taking special care to inject in the "corner pocket".
  Arms: Bupivacaine HCL plus supraclavicular block
Drug: Group C(supraclavicular block only) — In the recovery room the patient will be given the supraclavicular block which will be ultrasound guided and consisting of 20 cc of Bupivacaine HCl 0.25% .Anesthesiologist performing the block will be instructed to surround the brachial plexus with the local anesthetic, taking special care to inject in the "corner pocket".
  Arms: supraclavicular block only

SUMMARY:
The purpose of this study is to see if Exparel, used intraoperatively by injecting at the surgical site, followed by a Supraclavicular nerve block with bupivacaine in the recovery room, will provide better pain scores for patients at 24 and 48 hours post operatively than, 1)Bupivacaine Hydrochloride (HCL) injection at the surgical site, with a supraclavicular block in Post-anesthesia care unit(PACU), or 2)a supraclavicular block in PACU without any kind of injection at the surgical site.

ELIGIBILITY:
Inclusion Criteria:

* distal radius fractures
* undergoing Open reduction internal fixation (ORIF) at Lyndon B Johnson Ambulatory Surgical Center (LBJ ASC)

Exclusion Criteria:

* pregnancy
* history of chronic pain conditions
* currently taking opioids

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2021-11-20 (Estimated); Study Completion 2021-11-20 (Estimated)

PRIMARY OUTCOMES:
Pain as measured by the Revised American Pain Society Patient Outcome Questionnaire (APS-POQ-R) | 24 hours post treatment
  The questionnaire consists of 13 questions.The first 11 is scored form 0-10(a higher number indicating a worse outcome).
Pain as measured by the Revised American Pain Society Patient Outcome Questionnaire (APS-POQ-R) | 48 hours post treatment
  The questionnaire consists of 13 questions.The first 11 is scored form 0-10(a higher number indicating a worse outcome).

SECONDARY OUTCOMES:
Number of patients who presented to Emergency room following surgery for pain control | 24 hours post surgery
Number of patients who presented to Emergency room following surgery for pain control | 48 hours post surgery
Number of over the counter(OTC) pain medications consumed by the patient | 24 hours post surgery
Number of OTC pain medications consumed by the patient | 48 hours post surgery
Number of prescription opioid medications consumed by the patient | 24 hours post surgery
Number of prescription opioid medications consumed by the patient | 48 hours post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Erikka L Washington, MD, Principal Investigator — The University of Texas Health Science Center, Houston

IPD SHARING:
Plan to Share IPD: No